CLINICAL TRIAL: NCT00740857
Title: A Study Comparing the Efficacy of Two Ibuprofen Formulations
Brief Title: Study Comparing the Efficacy of Two Ibuprofen Formulations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PV-08-24
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2010-08-12 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2011-06

CONDITIONS: Pain
Keywords: Dental pain analgesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Active Comparator)
  Interventions: Drug: ibuprofen Formulation 1
- 3 (Active Comparator)
  Interventions: Drug: ibuprofen Formulation 2

INTERVENTIONS:
Drug: placebo — 2 placebo gels capsules delivered as a single dose.
  Arms: 1
Drug: ibuprofen Formulation 1 — 2 marketed ibuprofen gels
  Arms: 2
Drug: ibuprofen Formulation 2 — 2 marketed ibuprofen gels
  Arms: 3

SUMMARY:
This is a study of healthy volunteers to compare how quickly different ibuprofen products relieve dental pain.

ELIGIBILITY:
Inclusion criteria :

* Outpatients with post-operative pain following surgical extraction of third molars,
* examined by the attending dentist or physician and medically cleared to participate in the study,
* in general good health and have no contraindications to the study or rescue medication.

Exclusions criteria:

* any serious medical condition,
* acute localized dental infection at the time of surgery ,
* females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years and not using a medically approved method of contraception.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 211 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the United States from August 2008 to October 2008.
Pre-assignment Details: During the screening period, the Investigator or his/her designee examined each subject and completed a checklist of the inclusion/exclusion criteria in order to determine the patient's eligibility. Surgery occurred within 14 days of the screening visit.
Groups:
- Placebo: 2 placebo gel capsules delivered as a single dose up to 5 hours after surgery
- Ibuprofen Formulation 1: 2 marketed ibuprofen 200 mg liquid gels up to 5 hours after surgery
- Ibuprofen Formulation 2: 2 marketed ibuprofen 200 mg soft gels up to 5 hours after surgery
Period: Overall Study
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Started | 33 | 88 | 90
Completed | 32 | 88 | 90
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2 | Total
Number analyzed (Participants) | 33 | 88 | 90 | 211
Age Continuous [Mean (Standard Deviation); unit: years] | 18.8 (2.7) | 18.5 (2.5) | 19.0 (3.0) | 18.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 43 | 45 | 104
  Male | 17 | 45 | 45 | 107

OUTCOME MEASURES:

1. Primary Outcome: Time to Meaningful Pain Relief
Description: Subjects evaluated the time to "First Perceptible" Relief by depressing a stopwatch at the moment they first began to experience "perceptible" relief and the time to "Meaningful" Relief by depressing a second stopwatch at the moment they first began to experience "meaningful" relief. These times were recorded up to 6 hrs after dosing. Range: up to 6 hrs, a lower number is better.
Time Frame: 0-6 hours
Population: All randomized patients who were dosed with study product, indicated a baseline score of at least 2 out of 4 on the Categorical Pain Severity Rating Scale and confirmed a pain assessment of at least 50 mm out of 100 mm on the Visual Analog Scale (VAS). Median pain relief was not reached for the placebo participants within 360 minutes.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 0 | 88 | 90
minutes |  | 45.4 [41.5 to 53.5] | 63.6 [58.6 to 84.0]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms
Statistical Analysis 2: Comparison: Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; Test type: Superiority or Other; p = 0.001, Proportional hazards model; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Formulation 2; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms

2. Secondary Outcome: Pain Intensity Difference (PID) Scores at Each Individual Time Points
Description: PID is based on the 4-point categorical pain severity score ranging from 0 (none) to 3 (severe), this value was derived by subtracting the score at each post-dosing time point from the baseline score, so that a higher positive value is indicative of greater improvement.
Time Frame: 0-6 hours
Population: All randomized patients who were dosed with study product, indicated a baseline score of at least 2 out of 4 on the Categorical Pain Severity Rating Scale and confirmed a pain assessment of at least 50 mm out of 100 mm on the Visual Analog Scale (VAS).
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 33 | 88 | 90
units on scale
  15 minutes | 0.1 (0.4) | 0.2 (0.5) | 0.1 (0.3)
  30 minutes | 0.2 (0.5) | 0.8 (0.8) | 0.5 (0.6)
  45 minutes | 0.3 (0.7) | 1.3 (0.8) | 0.9 (0.7)
  60 minutes | 0.3 (0.7) | 1.6 (0.9) | 1.2 (0.8)
  90 minutes | 0.2 (0.8) | 1.8 (0.9) | 1.5 (0.8)
  120 minutes | 0.2 (0.8) | 1.8 (0.9) | 1.7 (0.8)
  180 minutes | 0.3 (1.0) | 1.7 (1.0) | 1.7 (0.9)
  240 minutes | 0.4 (1.2) | 1.5 (1.0) | 1.5 (0.9)
  300 minutes | 0.2 (1.0) | 1.4 (1.0) | 1.4 (1.0)
  360 minutes | 0.2 (1.0) | 1.2 (1.0) | 1.3 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; 15 minutes; Test type: Superiority or Other; p = 0.118, ANOVA; With treatment, baseline Pain Severity Rating (PSR), and gender terms
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; The 30, 45, 60; Test type: Superiority or Other; p < 0.001, ANOVA; With treatment, baseline Pain Severity Rating (PSR), and gender terms

3. Secondary Outcome: Pain Relief (PR) Scores at Individual Time Points
Description: Response to the question "How much pain do you have from your starting pain?" was recorded on a 5-point categorical pain relief scale (None (0), A Little (1), Some (2), A Lot (3) or Complete (4)) at designated time points after study medication was taken.
Time Frame: 0-6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 33 | 88 | 90
units on scale
  15 minutes | 0.2 (0.5) | 0.5 (0.8) | 0.3 (0.6)
  30 minutes | 0.6 (0.8) | 1.6 (1.1) | 1.0 (0.9)
  45 minutes | 0.8 (1.0) | 2.4 (1.1) | 1.7 (1.1)
  60 minutes | 0.9 (1.1) | 2.9 (1.0) | 2.1 (1.1)
  90 minutes | 0.8 (1.1) | 3.2 (1.0) | 2.7 (1.0)
  120 minutes | 0.8 (1.2) | 3.2 (1.0) | 2.9 (1.0)
  180 minutes | 1.0 (1.4) | 3.0 (1.1) | 2.9 (1.1)
  240 minutes | 1.1 (1.6) | 2.7 (1.2) | 2.7 (1.2)
  300 minutes | 0.8 (1.2) | 2.5 (1.4) | 2.6 (1.3)
  360 minutes | 0.8 (1.3) | 2.2 (1.3) | 2.6 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; 15 minutes; Test type: Superiority or Other; p = 0.041, ANOVA; With treatment, baseline Pain Severity Rating (PSR), and gender terms
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; The 30, 45, 60, 90, 120, 180, 240, 300 and 360 minute individual time points all have the same P-value score; Test type: Superiority or Other; p < 0.001, ANOVA; With treatment, baseline Pain Severity Rating (PSR), and gender terms

4. Secondary Outcome: Time-weighted Sum of Pain Relief + Pain Intensity Difference (SPRID) From 0-2 Hours and 0-6 Hours
Description: SPRID is a derived endpoint from the pain relief and pain intensity difference scores from 0-2 hours and 0-6 hours. PRID=PID+Pain Relief Score. SPRID-02 range: -2 (worst) to 14 (best); SPRID 06 range: -6 (worst) to 42 (best).
Time Frame: 0-2 and 0-6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 33 | 88 | 90
units on scale
  0-2 hours | 1.8 (2.9) | 7.8 (2.9) | 6.3 (2.6)
  0-6 hours | 6.5 (11.9) | 24.0 (10.1) | 23.0 (9.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; Test type: Superiority or Other; p < 0.001, ANOVA; With treatment, baseline Pain Severity Rating (PSR), and gender terms

5. Secondary Outcome: Pain Relief Combined With Pain Intensity Difference (PRID) Scores at Individual Time Points
Description: PRID (PRID=PID+PR) is a derived endpoint from the pain relief and pain intensity difference scores at each time point. Range: -1 (worst) to 7 (best).
Time Frame: 0-6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 33 | 88 | 90
units on scale
  15 minutes | 0.3 (0.8) | 0.7 (1.2) | 0.4 (0.9)
  30 minutes | 0.8 (1.2) | 2.4 (1.8) | 1.4 (1.5)
  45 minutes | 1.1 (1.6) | 3.6 (1.8) | 2.5 (1.7)
  60 minutes | 1.2 (1.8) | 4.5 (1.8) | 3.3 (1.7)
  90 minutes | 1.0 (1.9) | 5.0 (1.7) | 4.2 (1.7)
  120 minutes | 1.0 (2.0) | 5.0 (1.8) | 4.6 (1.7)
  180 minutes | 1.2 (2.4) | 4.7 (2.0) | 4.6 (1.8)
  240 minutes | 1.5 (2.7) | 4.2 (2.1) | 4.2 (2.0)
  300 minutes | 1.0 (2.1) | 3.9 (2.3) | 4.0 (2.2)
  360 minutes | 1.0 (2.2) | 3.4 (2.3) | 3.9 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; 15 minutes; Test type: Superiority or Other; p = 0.056, ANOVA; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; The 30, 45, 60, 90, 120, 180, 240, 300 and 360 minute individual time points all have the same P-value score; Test type: Superiority or Other; p < 0.001, ANOVA; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms

6. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference (SPID) From 0-2 Hours and 0-6 Hours
Description: SPID is a derived endpoint from the pain intensity difference scores from 0-2 hours and 0-6 hours. Range: -2 (worst) to 6 (best); -6 (worst) to 18 (best).
Time Frame: 0-2 and 0-6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 33 | 88 | 90
units on scale
  0-2 hours | 0.4 (1.2) | 2.8 (1.4) | 2.2 (1.1)
  0-6 hours | 1.4 (5.2) | 8.6 (4.8) | 8.1 (4.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; Test type: Superiority or Other; p < 0.001, ANOVA; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms

7. Secondary Outcome: Time-weighted Sum of Pain Relief Scores (TOTPAR) From 0-2 Hours and 0-6 Hours
Description: TOTPAR is a derived endpoint from the pain relief scores from 0-2 hours and 0-6 hours. Range: 0 (worst) - 8 (best); 0 (worst) - 24 (best)
Time Frame: 0-2 and 0-6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 33 | 88 | 90
units on scale
  0-2 hours | 1.4 (1.8) | 5.0 (1.7) | 4.1 (1.6)
  0-6 hours | 5.1 (7.1) | 15.4 (5.7) | 14.9 (5.8)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; Test type: Superiority or Other; p < 0.001, ANOVA; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms

8. Secondary Outcome: Time to First Perceptible Relief
Description: The elapsed time from dosing until the patient indicated first perceptible relief, provided the subject also indicated achieving meaningful relief.
Time Frame: 0-6 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Number analyzed (Participants) | 0 | 88 | 90
minutes |  | 23.7 [20.6 to 26.6] | 28.6 [25.9 to 31.5]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Formulation 1 vs Ibuprofen Formulation 2; Test type: Superiority or Other; p < 0.001, proportional hazards model; Adjusted with treatment, baseline Pain Severity Rating (PSR), and gender terms

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen Formulation 1 | Ibuprofen Formulation 2
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/88 | 0/90
Other Adverse Events (participants affected / at risk) | 13/33 | 2/88 | 7/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=33) | Ibuprofen Formulation 1 (N=88) | Ibuprofen Formulation 2 (N=90)
Nausea (Gastrointestinal disorders) | 4 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0
Dry socket (Infections and infestations) | 0 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agreed to allow the sponsor 30 days to review and approve abstracts and 60 days to review and approve manuscripts prior to submission to protect against disclosure of confidential information.